CLINICAL TRIAL: NCT01125696
Title: Maternal Tenofovir-containing Combination Drug Regimen During the Second and Third Trimesters of Pregnancy for Prevention of Mother-to-child Transmission of HIV and HBV in HIV-HBV Co-infected Mothers
Brief Title: Safety Study of a Tenofovir-containing Drug Regimen for the Prevention of Mother-to-child Transmission of HIV and HBV
Acronym: TiP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: National Center for AIDS/STD Control and Prevention, China CDC (Other Government)
Responsible Party: Principal Investigator, Athena Kourtis, Lead Medical Officer, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCCDPHP-5877
Record Dates: First submitted 2010-03-29; First posted 2010-05-18 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: HIV; Hepatitis B
Keywords: mother-to-child transmission; HIV; Hepatitis B; Pregnant women; Tenofovir; Infants
MeSH Terms: conditions — Hepatitis B | interventions — Tenofovir; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard of Care (Active Comparator)
  Interventions: Drug: Zidovudine/lamivudine/lopinavir-ritonavir
- Tenofovir (Experimental)
  Interventions: Drug: Tenofovir/lamivudine/lopinavir-ritonavir

INTERVENTIONS:
Drug: Tenofovir/lamivudine/lopinavir-ritonavir — Tenofovir/lamivudine/lopinavir-ritonavir given to mothers starting at 14-28 weeks gestation till labor/delivery and continued postpartum if maternal baseline CD4<350
  Arms: Tenofovir
Drug: Zidovudine/lamivudine/lopinavir-ritonavir — Zidovudine/lamivudine/lopinavir-ritonavir given to mothers starting at 14-28 weeks gestation till labor/delivery and continued postpartum if maternal baseline CD4<350
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to compare a regimen of tenofovir/lamivudine/lopinavir-ritonavir to the WHO-recommended and locally practiced standard of care regimen consisting of zidovudine/lamivudine/lopinavir-ritonavir during the second and third trimesters of pregnancy in HIV and HBV co-infected women. This is a phase II study evaluating the safety of the test regimen in pregnant women and their newborns. While the study is not powered to examine efficacy, preliminary estimates of transmission of HIV and HBV to the infants and of the rate of resistance development will be obtained.

DETAILED DESCRIPTION:
Great progress has been made in preventing mother-to-child transmission (MTCT) of HIV in resource-rich settings with the use of combination antiretroviral regimens during pregnancy and peripartum. In the resource-limited world simple inexpensive regimens administered peripartum, such as single dose nevirapine to mothers and infants, have been effective in reducing transmission but at the cost of development of resistance. Strategies that will allow women to preserve their antiretroviral options when they will need therapy for their own HIV disease and will improve efficacy are urgently needed. Moreover, co-infection with hepatitis B virus (HBV) is a problem for a substantial proportion of HIV-infected pregnant women. HIV alters the course of HBV disease by increasing levels of HBV DNA replication and thus risk of transmission to the newborn. HBV immunization in the infant with the first dose started soon after birth has decreased the bulk of such transmission, but the risk remains, particularly for mothers with HBe antigen positivity. Ideally an antiviral regimen administered during pregnancy with activity against both viruses would minimize transmission of both HIV and HBV to the infant.

The investigators propose to study a combination of tenofovir/lamivudine/lopinavir-ritonavir started between 14 and 28 weeks of pregnancy in HIV and HBV co-infected women. This regimen provides potent antiviral activity for prevention of MTCT. In addition, tenofovir and lamivudine both have activity against HBV, and could play a role in decreasing transmission of HBV to the infant. This regimen will be compared to the WHO-recommended and locally practiced standard of care, consisting of zidovudine/lamivudine/lopinavir-ritonavir, also starting at 14-28 weeks of pregnancy. This will be a phase II study evaluating the safety of the test regimen in pregnant women and their newborns, in particular renal, bone mineral density and hepatic toxicity (including hepatic flares post discontinuation of therapy). The study will recruit 80 pregnant women of at least 20 years of age in China and follow them and their infants for 12 months post-delivery. The investigators will recruit from prenatal clinics in some of the districts most heavily affected by HIV in the Guangxi province in China. China is selected for this study as it is hyperendemic for hepatitis B and has a rising HIV epidemic. Although not powered to examine efficacy, preliminary estimates of transmission of HIV and HBV to the infants and of the rate of resistance development will be obtained. The study will be done in collaboration with CDC-GAP China and the Chinese Ministry of Health-National Center for AIDS, which will coordinate recruitment, study visits and data collection through the local HIV/AIDS coordinators.

ELIGIBILITY:
Inclusion Criteria:

* Serologically-confirmed HIV and HBV infection
* Gestational age less than 28 weeks
* Willingness to participate in a clinical trial
* Age 20 years or over on the day of inclusion
* Willingness to return for follow-up visits and to allow infant participation in the trial
* Intent to remain in the clinic catchment area during the duration of the study
* No serious current complications of pregnancy
* No previous or current use of antiretrovirals including the HIVNET 012 regiment
* Hemoglobin over 8 g/dL
* Blood creatinine clearance greater than or equal to 60 mL/min estimated by the Cockroft-Gault formula for women

Exclusion Criteria:

* Age less than 20
* Pregnant woman refuses to sign the consent to participate
* Unwillingness to adhere to visit schedule or maintain adherence with medications
* Illnesses so severe as to likely require maternal hospitalization
* Intend to breastfeed

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-05; Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Tenofovir Safety for mothers measured by incidence of serious adverse events (SAEs) | From baseline (14-28 weeks gestation) through 12 months postpartum
  SAEs will be defined using the DAIDS Toxicity Tables
Dual Energy X-ray absorptiometry (DXA) scans of bone mineral density | from delivery through 6 months postpartum
  Mothers will have DXA scan of hip and lumbar spine. Infants will have DXA scan of whole body and lumbar spine.
Maternal Tenofovir Pharmacokinetics | 16 weeks gestation through delivery
  Only for mothers on the active arm.
Infant Tenofovir Pharmacokinetics | one timepoint within 12 hours of delivery
  Only for infants on the active arm.
Tenofovir safety for infants measured by incidence of serious adverse events (SAEs) | from birth through 12 months of age
  SAEs defined according to the DAIDS toxicity tables.

SECONDARY OUTCOMES:
HBV viral load in mothers | from baseline (14-28 weeks gestation) through delivery
Infant HIV transmission rate | birth through 12 months
Infant HBV transmission rate | birth through 12 months
Prevalence of HIV resistance mutations | from baseline (14-28 weeks gestation) through 12 months postpartum
Prevalence of HBV resistance mutations | from baseline (14-28 weeks gestation) through 12 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Athena P Kourtis, MD, PhD, MPH, Principal Investigator — Centers for Disease Control and Prevention, Division of Reproductive Health
Locations (2):
- China (2):
  - Liuzhou MCH Hospital, Liuchow, Guangxi
  - Guangxi MCH Hospital, Nanning, Guangxi

REFERENCES:
- [Derived] Wang L, Wiener J, Bulterys M, Wei X, Chen L, Liu W, Liang S, Shepard C, Wang L, Wang A, Zhang F, Kourtis AP. Hepatitis B Virus (HBV) Load Response to 2 Antiviral Regimens, Tenofovir/Lamivudine and Lamivudine, in HIV/ HBV-Coinfected Pregnant Women in Guangxi, China: The Tenofovir in Pregnancy (TiP) Study. J Infect Dis. 2016 Dec 1;214(11):1695-1699. doi: 10.1093/infdis/jiw439. Epub 2016 Sep 22. PMID 27658693